CLINICAL TRIAL: NCT04314791
Title: Accuracy of Placenta Accreta Index in Diagnosing Placenta Accreta Spectrum: A Prospective Study
Brief Title: Accuracy of Placenta Accreta Index in Diagnosing Placenta Accreta Spectrum
Status: Completed | Type: Observational
Sponsor: Hatem AbuHashim (Other)
Responsible Party: Sponsor-Investigator, Hatem AbuHashim, Professor, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: MS.17.04.143
Record Dates: First submitted 2020-03-14; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- US scan with calculation of the PAI
  Interventions: Device: Ultrasound evaluation, with grayscale and color Doppler imaging

INTERVENTIONS:
Device: Ultrasound evaluation, with grayscale and color Doppler imaging — In pregnant women with previous CS and anterior low-lying or placenta previa, the following three sonographic criteria were assessed: (i) the smallest myometrial thickness in the sagittal plane; (ii) presence of placental lacunae and its grade from 0-3; (iii) bridging vessels using color Doppler. The PAI score (up to 9) was calculated for every patient as described by Rac et al.2015.

SUMMARY:
The placenta accreta spectrum (PAS) which includes accreta, increta, and percreta represents a significant obstetric challenge. PAS complicates as many as 1 per 500 pregnancies and this risk is increased with prior cesarean deliveries. Antenatal diagnosis of PAS allows for multidisciplinary planning and delivery before the onset of labor and/or vaginal bleeding. This approach has reduced maternal morbidity rates, including less blood loss, fewer transfusion requirements and, intraoperative urologic injuries as well as improve fetal outcome.

Ultrasound evaluation, with grayscale and color Doppler imaging, is the recommended first-line modality for diagnosing PAS. Grayscale ultrasound features suggestive of placenta accreta include an inability to visualize the normal retroplacental clear zone, irregularity, and attenuation of the uterine-bladder interface, retroplacental myometrial thickness, presence of intraplacental lacunar spaces, and bridging vessels between the placenta and bladder wall when using color Doppler.

The placenta accreta index (PAI) score (a nine-point score) was proposed in 2015 to predict PAS based on US parameters in a high-risk population by retrospective data analysis. The probability of histological invasion was found to increase with increasing the PAI score. This study aimed to prospectively evaluate the diagnostic performance of the PAI in the prediction of PAS in relation to histopathological findings.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their third trimester
* with a single fetus in the current pregnancy
* a previous delivery by at least 1 cesarean section
* having an anterior placenta previa or anterior low-lying placenta by ultrasound assessment

Exclusion Criteria:

* cases with twin or multiple pregnancies,
* cases with a non-previa placenta or posterior low lying or previa placenta,
* cases without previous deliveries by cesarean section
* cases before the third trimester of pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant females during the third trimester of pregnancy, with a single fetus in the current pregnancy, a previous delivery by at least 1 cesarean section and having an anterior placenta previa or anterior low-lying placenta by ultrasound assessment.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the PAI | through study completion, an average of 1 year
  The diagnostic accuracy of the PAI in comparison with the histopathological confirmation in hysterectomy specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, Study Chair — Faculty of Medicine, Mansoura University; Eman Shalaby, Principal Investigator — Mansoura University Hospital
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Background] Rac MW, Dashe JS, Wells CE, Moschos E, McIntire DD, Twickler DM. Ultrasound predictors of placental invasion: the Placenta Accreta Index. Am J Obstet Gynecol. 2015 Mar;212(3):343.e1-7. doi: 10.1016/j.ajog.2014.10.022. Epub 2014 Oct 18. PMID 25446658